CLINICAL TRIAL: NCT05716841
Title: Effects of Ballistic Exercises on Pain, Disability, and Explosive Strength in Tennis Players With Shoulder Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Usama sohail0439
Record Dates: First submitted 2023-01-18; First posted 2023-02-08 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): It was treated with stretching and simple baseline strengthening of the upper limb through any regular mean (like TheraBand) in a moderate manner with 10 to 20 repetitions for 3 days per week for six weeks.
- Experimental group (Experimental): This experimental group was treated with stretching and then strengthening of the upper limb through ballistic six exercises from a moderate to intense manner with 3 sets of 10 repetitions with a 30 sec gap between sets, 3 sets of 15 repetitions with a 30sec gap between sets, and 3 sets of 20 repetitions with a 30sec gap between sets for 3 to 4 days per week for six weeks.
  Interventions: Other: Ballistic exercises

INTERVENTIONS:
Other: Ballistic exercises — stretching and then strengthening of the upper limb through ballistic six exercises from a moderate to intense manner with 3 sets of 10 repetitions with a 30sec gap between sets, 3 Sets of 15 repetitions with a 30sec gap between sets, and 3 sets of 20 repetitions with a 30sec gap between sets for 3 to 4 days per week for six weeks.
  Arms: Experimental group

SUMMARY:
The goal of this Randomized control trial is to determine ''Effects of ballistic exercises on pain, disability and explosive strength in tennis players with shoulder pain''. The main question it aims to answer is:

To determine effect of ballistic exercises on pain, disability and explosive strength in tennis players with shoulder pain.

Participants will be divided into 2 groups. Group-A will be treated with stretching and simple baseline strengthening of the upper limb through any regular mean (like TheraBand) in a moderate manner with 10 to 20 repetitions for 3 days per week for six weeks. Group B will be treated with stretching and then strengthening of the upper limb through ballistic six exercises from a moderate to intense manner with 3 sets of 10 repetitions with a 30sec gap between sets, 3 sets of 15 repetitions with a 30sec gap between sets, and 3 sets of 20 repetitions with a 30sec gap between sets for 3 to 4 days per week for six weeks.

DETAILED DESCRIPTION:
Sporting events that necessitate the regular use of an upper limb necessitate the highest kinetic chain efficiency in this section. Dysfunction of the musculoskeletal system, coupled with failure in motor abilities, might expose adolescents to significant complaints of chronic conditions, especially for the shoulder.

Tennis players are prone to shoulder discomfort and injury. The particular reasons for such discomfort are unknown. Impingement at significant tennis positions and glenohumeral instability has never been examined in vivo dynamically. Injuries of the rotator cuff are a major source of discomfort and dysfunction among tennis players and other overhead athletes. The etiology of rotator cuff tears in tennis players is multifaceted, with microtrauma and internal impingement causing partial tears in younger athletes and degenerative full-thickness tears in older players

The goal of this Randomized control trial is to determine ''Effects of ballistic exercises on pain, disability and explosive strength in tennis players with shoulder pain''. The main question it aims to answer is:

To determine effect of ballistic exercises on pain, disability and explosive strength in tennis players with shoulder pain.

Participants will be divided into 2 groups. Group-A will be treated with stretching and simple baseline strengthening of the upper limb through any regular mean (like TheraBand) in a moderate manner with 10 to 20 repetitions for 3 days per week for six weeks. Group B will be treated with stretching and then strengthening of the upper limb through ballistic six exercises from a moderate to intense manner with 3 sets of 10 repetitions with a 30sec gap between sets, 3 sets of 15 repetitions with a 30sec gap between sets, and 3 sets of 20 repetitions with a 30sec gap between sets for 3 to 4 days per week for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age will be 18 to 35 years.
* Gender: Both Male and Female.
* Players playing on a regular basis will be targeted in this study.
* Players with upper limb disability with Quick DASH Score of more than 6 percent.

Exclusion Criteria

* History of any neurological impairment as described by the player which may affect the outcome of the study.
* Any history of the pathological status of bones or joints as described by the player which may affect the outcome of a study
* Any history of musculoskeletal or traumatic status as described by the player which may affect the outcome of the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Push-ups and Pull ups test (for shoulder strength) | 6 weeks
  The push-up fitness test (also called the press-up test) measures upper body strength and endurance. There are many variations of the push-up test, with differences in the placement of the hands, how far to dip, the duration of the test, and the method of counting the number of completed push-ups. Here we discuss the general method for the push-up test and link to specific push-up fitness tests. Its reliability is 0.93.
Numeric Pain Rating scale | 6 weeks
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Quick DASH Questionaries | 6 weeks
  The purpose of the Quick DASH is to use 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. The Quick DASH is a widely used reference for self-reported disability.

CONTACTS AND LOCATIONS:
Overall Officials: Usama Sohail, MSPT, Principal Investigator — Riphah International University, Lahore
Locations (1):
- Pakistan sports board and coaching center, Lahore, Punjab Province, Pakistan